CLINICAL TRIAL: NCT01553539
Title: A Phase II Clinical Trial of Angiotensin 1-7 For the Second or Third Line Treatment of Patients With Metastatic or Unresectable Sarcomas
Brief Title: Therapeutic Angiotensin-(1-7) in Treating Patients With Metastatic Sarcoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00008212; NCI-2009-01259 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 003936-01A2 (Other Grant/Funding Number: FDA OOPD); CCCWFU 71108 (Other: Wake Forest University Health Sciences); NCT00974545 (obsolete NCT alias)
Record Dates: First submitted 2012-03-09; First posted 2012-03-14 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Bone Cancer; Chondrosarcoma; Clear Cell Sarcoma of the Kidney; Metastatic Osteosarcoma; Ovarian Sarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Osteosarcoma; Recurrent Uterine Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage III Uterine Sarcoma; Stage IV Adult Soft Tissue Sarcoma; Stage IV Uterine Sarcoma
MeSH Terms: conditions — Bone Neoplasms; Chondrosarcoma; Osteosarcoma; Sarcoma | interventions — angiotensin I (1-7)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (antiangiogenesis therapy) (Experimental): Patients receive therapeutic angiotensin-(1-7) SC once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: therapeutic angiotensin-(1-7); Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: therapeutic angiotensin-(1-7) — Given SC
  Other Names: therapeutic Ang-(1-7); TXA127
Other: laboratory biomarker analysis — Correlative study

SUMMARY:
This phase II trial studies how well therapeutic angiotensin-(1-7) works as second-line therapy or third-line therapy in treating patients with metastatic sarcoma that cannot be removed by surgery. Therapeutic angiotensin-(1-7) may stop the growth of sarcoma by blocking blood flow to the tumor.

Funding Source - FDA Office of Orphan Drug Products (OOPD)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate of chemotherapy-refractory sarcomas to 20 mg per day of single-agent Ang(Angiotensin)-(1-7) or 10 mg per day of single-agent Ang-(1-7) if excessive toxicity is observed at the 20 mg dose.

II. To evaluate toxicities associated with single-agent Ang-(1-7) when given to patients with chemotherapy-refractory sarcomas.

SECONDARY OBJECTIVES:

I. To assess time to progression (TTP) and overall survival (OS) in patients treated with Ang-(1-7).

II. To evaluate accumulation of Ang-(1-7) after 21 days of continuous treatment and quantify changes in plasma levels of angiogenic peptides including placental growth factor (PlGF).

OUTLINE:

Patients receive therapeutic angiotensin-(1-7) subcutaneously (SC) once daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed sarcoma that is metastatic or unresectable and have progressed despite 1 or 2 prior treatment regimens with chemotherapy or targeted anti-cancer agents such as imatinib
* Prior treatment: >= 4 weeks since completion of radiation or chemotherapy, except for >= 6 weeks for Melphalan, nitrosoureas, or mitomycin-C
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1,500/Microliter (mcL)
* Platelets >= 100,000/mcL
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) < 3 X upper limit or normal (ULN)
* Estimated (est.) creatinine clearance > 30 mL/min
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as > 10 mm
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or double-barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents for cancer treatment
* Patients with evidence of bleeding diathesis are ineligible
* No concurrent treatment with angiotensin-converting-enzyme (ACE) inhibitors or angiotensin II receptor blockers (ARBs)
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or hypotension, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and nursing women are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Petty, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Antiangiogenesis Therapy): Patients receive therapeutic angiotensin-(1-7) subcutaneous (SC) once daily in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Antiangiogenesis Therapy)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Activity as Assessed by Number of Patients Showing an Objective Tumor Response
Description: 'Activity' will be operationalized using objective tumor response, which will be estimated as the proportion of partial and complete responders (according to Response Evaluation Criteria in Solid Tumors [RECIST] criteria) among all evaluable patients. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Approximately 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 20
participants | 0

2. Primary Outcome: Number of Participants Who Experienced Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: See the adverse event tables for specifics.
Time Frame: Approximately 1 year
Measure: Number; unit: Participants experiencing adverse events
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 20
Participants experiencing adverse events | 20

3. Secondary Outcome: Time to Disease Progression
Time Frame: Approximately 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 20
months | 2.7 [1.4 to 4.1]

4. Secondary Outcome: Overall Survival
Time Frame: Approximately 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 20
months | 10.2 [5.3 to 18.3]

5. Secondary Outcome: Plasma Levels of Angiogenic Peptides Including Placental Growth Factor (PlGF)
Time Frame: Baseline and Day 22
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 20
pg/mL
  Ang-(1-7) Baseline | 18.4 (385.0)
  Ang-(1-7) Day 22 | 41.2 (2840.0)
  Ang II Baseline | 21.3 (11.5)
  Ang II Day 22 | 31.5 (26.5)
  Ang I Baseline | 22.5 (127)
  Ang I Day 22 | 17.5 (52.7)
  VEGF Baseline | 65.6 (66.4)
  VEGF Day 22 | 49.6 (43.0)
  PIGF Baseline | 4.3 (2.1)
  PIGF Day 22 | 3.0 (1.7)

ADVERSE EVENTS:
Time Frame: Duration of treatment, up to one year
Description: worst of each type of adverse event was recorded for each patient
Arm/Group | Treatment (Antiangiogenesis Therapy)
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antiangiogenesis Therapy) (N=20)
Low Hemoglobin (Investigations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hyperglycemia (Investigations) | 2 (2)
hypomagnesemia (Investigations) | 1 (1)
hyponatremia (Investigations) | 2 (2)
hypokalemia (Investigations) | 1 (1)
hypoalbuminemia (Investigations) | 2 (2)
hyperbilirubinemia (Investigations) | 1 (1)
serum glutamic pyruvic transaminase (Investigations) | 1 (1)
hypophosphatemia (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
serum glutamic oxaloacetic transaminase (Investigations) | 1 (1)
hyperkalemia (Investigations) | 1 (1)
Hypoxia (Investigations) | 2 (2)
hyperuricemia (Investigations) | 1 (1)
Pain: Abdomen (General disorders) | 2 (2)
Acidosis (Investigations) | 2 (2)
Alkalosis (Investigations) | 1 (1)
Pain: Chest wall (General disorders) | 1 (1)
Obstruction, GI: Colon (Gastrointestinal disorders) | 1 (1)
Lymphopenia (Investigations) | 4 (4)
Muscle weakness (General disorders) | 2 (2)
Pain: Extremity-limb (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Pain: Pleura (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Pain: Stomach (General disorders) | 1 (1)
Supraventricular and nodal arrhythmia: Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Obstruction, GU: Ureter (General disorders) | 3 (3)
Pain: Urethra (General disorders) | 1 (1)
Urinary with low grade neutropenia (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: Oral cavity-gums (Infections and infestations) | 1 (1)
Prolapse of stoma, GI (Gastrointestinal disorders) | 1 (1)
Infection Biliary tree (Infections and infestations) | 1 (1)
Infection with unknown ANC Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Intra-operative injury: Spinal cord (General disorders) | 1 (2)
Blood Infection with high grade neutropenia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antiangiogenesis Therapy) (N=20)
Creatinine (Investigations) | 2 (2)
Dizziness (General disorders) | 2 (2)
Taste alteration (General disorders) | 2 (2)
Bicarbonate serum-low (Investigations) | 2 (2)
hyperbilirubinemia (Investigations) | 2 (2)
serum glutamic pyruvic transaminase (Investigations) | 2 (2)
Pain: Head/headache (General disorders) | 2 (2)
hypermagnesemia (Investigations) | 2 (2)
Heartburn/dyspepsia (General disorders) | 2 (2)
Depression (General disorders) | 2 (2)
Muscle weakness (General disorders) | 2 (2)
Pain: Muscle (General disorders) | 2 (2)
Pain: Dental/teeth/peridontal (General disorders) | 2 (2)
Urinary retention (including neurogenic bladder) (General disorders) | 3 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypotension (Cardiac disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Sweating (General disorders) | 3 (3)
hypocalcemia (Investigations) | 3 (3)
serum glutamic oxaloacetic transaminase (Investigations) | 3 (3)
Dehydration (General disorders) | 3 (3)
Anxiety (General disorders) | 3 (3)
Partial Thromboplastin Time (Investigations) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pain: Chest/thorax (General disorders) | 3 (3)
Pain: Neck (General disorders) | 3 (3)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 3 (3)
Hemorrhage pulmonary/upper respiratory (Vascular disorders) | 3 (3)
Insomnia (General disorders) | 4 (4)
Weight loss (General disorders) | 4 (4)
Pruritus/itching (General disorders) | 4 (5)
Pain: Abdomen (General disorders) | 4 (4)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (5)
Proteinuria (Investigations) | 5 (5)
Neuropathy: sensory (Cardiac disorders) | 5 (5)
hyponatremia (Investigations) | 5 (5)
hypoalbuminemia (Investigations) | 5 (5)
Pain: Back (General disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Injection site reaction (Immune system disorders) | 6 (6)
low Platelets (Investigations) | 7 (7)
Anorexia (General disorders) | 7 (7)
Alkaline phosphatase (Investigations) | 7 (7)
Constipation (Gastrointestinal disorders) | 7 (7)
Pain: Joint (General disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 8 (8)
Fatigue (General disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Low WBC (Investigations) | 9 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
hypokalemia (Investigations) | 9 (9)
Edema: limb (Vascular disorders) | 9 (9)
Lymphopenia (Investigations) | 12 (12)
Low Hemoglobin (Investigations) | 14 (14)
hyperglycemia (Investigations) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes